CLINICAL TRIAL: NCT07149896
Title: A Prospective Randomized Controlled Study Of Collagen Scaffold For The Repair Of Elbow Cartilage Injury
Brief Title: A Study of Collagen Scaffold for the Repair of Elbow Cartilage Injury
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Chief physician, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K20250509-02
Record Dates: First submitted 2025-07-23; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cartilage Defect; Elbow Injury
Keywords: elbow cartilage defect; collagen scaffold
MeSH Terms: conditions — Elbow Injuries | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microfracture + Collagen scaffold (Experimental): After performing arthroscopic microfracture (with a cone tip spacing of 2-3mm and a depth reaching the subchondral bone), the defect site is dried using a suction tube and cotton swabs. A double-chamber syringe is used to inject the collagen scaffold, which will be then shaped and cured. Afterward, physiological saline is reinfused, and the stability of the graft is assessed under arthroscopy during the full range of motion of the elbow joint.
  Interventions: Device: Collagen Scaffold (Colla-Plug); Procedure: microfracture
- Microfracture (Active Comparator): Conventional arthroscopic microfracture operation is carried out, and the operation process of the experimental group is simulated by simulated drying and lavage during the operation.
  Interventions: Procedure: microfracture

INTERVENTIONS:
Device: Collagen Scaffold (Colla-Plug) — The collagen cartilage scaffold(COLTRIX® CartiRegen) used in this study consist of an injection needle, a syringe, and a collagen gel prefilled in a syringe. The collagen gel contains phosphate buffer and type Ⅰ collagen which the telopeptides are removed.. After the product is implanted in the body, it forms a degradable three-dimensional scaffold to provide an environment for cells to adhere, proliferate, migrate, differentiate and secrete, thereby promoting cartilage repair. At present, it has been commercially applied to clinical repair of knee cartilage defect.
  Arms: Microfracture + Collagen scaffold
Procedure: microfracture — Microfracture to repair cartilage defect is a minimally invasive procedure that is usually done arthroscopically. The doctor first cleans the damaged cartilage area, and then uses a special microfracture cone to drill vertically in the subchondral bone plate, forming multiple tiny holes, allowing mesenchymal stem cells and growth factors in the bone marrow to overflow, forming a blood clot rich in repair components, and finally stimulating fibrocartilage regeneration to fill the defect area.

SUMMARY:
The goal of this clinical trial is to test whether adding a collagen protein scaffold can improve cartilage repair in elbow joint injuries, compared to standard surgery alone. The study will enroll 90 patients (aged 18-55) with elbow cartilage damage who haven't responded to conservative treatments.

The main questions it aims to answer are:

* Does the collagen scaffold help regenerate better-quality cartilage (measured by MRI scans at 3 and 6 months)?
* Do patients experience better pain relief and elbow function after this combined treatment?

Researchers will compare two groups:

* Experimental group : Receives microfracture surgery + collagen scaffold implant
* Active Comparator group : Receives microfracture surgery alone

Participants will:

* Undergo arthroscopic surgery (either procedure)
* Complete follow-up visits at 1 week, 1 month, 3 months, and 6 months
* Have MRI scans and functional assessments
* Report pain levels and daily activity limitations through questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are between the ages of 18 and 55 (including 18 and 55 years old);
2. Articular cartilage defect reaches Outerbridge grade III/IV;
3. The area of cartilage defect in a single site is 0.5cm²-2cm²;
4. BMI 18≤BMI≤30;
5. Clinically diagnosed cartilage defect requiring arthroscopic microfracture;
6. Have not participated in other clinical trials within 3 months;
7. Conservative treatment such as rest/topical/oral non-steroidal anti-inflammatory drugs for more than 3 months has not been effective
8. Subjects fully understand the benefits and risks of this trial, are willing to participate and sign the informed consent form, and are able to cooperate with clinical follow-up.

Exclusion Criteria:

1. Obvious narrowing of the elbow joint space or bone ankylosis formed between joints;
2. Severe subchondral bone injury that cannot be undergoing microfracture surgery;
3. Those with severe elbow deformity or systemic osteoarticular diseases;
4. Secondary elbow arthritis with psoriasis, syphilitic neuropathy, brown yellow disease, metabolic bone disease;
5. Elbow joint cartilage damage caused by joint fractures, infections, tumors, and immune diseases;
6. Elbow joint tumors, rheumatoid, tuberculosis, suppuration and complications affecting the joint structure;
7. Those who have undergone cartilage defect transplantation from bone marrow mesenchymal stem cell transplantation or other cartilage regeneration surgery within 12 months before surgery;
8. Allergies, such as porcine protein allergy, past history or family history of autoimmune diseases;
9. Those who regularly use sedatives, sleeping pills, tranquilizers or other addictive drugs;
10. Combined with cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary diseases, mental illness;
11. Those who cannot receive long-term and complex rehabilitation training after surgery;
12. Women who are planning to have children, breastfeeding and pregnant women within 12 months;
13. Those who have contraindications to MRI examination;
14. Those who have special beliefs and cannot accept it (the product source is pig source);
15. Those who are not suitable for inclusion by other researchers, such as those who cannot be judged for efficacy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
MOCART(Magnetic Resonance Observation of Cartilage Repair Tissue) score | Preoperatively, 3rd and 6th months postoperatively
  The MOCART scoring system is a standardized assessment tool based on magnetic resonance imaging (MRI) specifically designed to quantify the morphological effects after articular cartilage repair. The scoring system uses a 100-point system (minimum score of 0, maximum score of 100), with higher scores representing better repair results. A total score of ≥75 indicates that the repaired tissue is close to normal hyaline cartilage in terms of structure, integration, and signal strength, while a score below 50 indicates poor repair effect or risk of complications. The assessment covered seven core indicators: volume filling of cartilage defects (0-20), integration with adjacent cartilage margins (0-15), repaired tissue surface structure (0-10), repaired tissue structure (0-10), repaired tissue signal intensity (0-15), subchondral bone changes (0-20), and bone quality changes (0-10).

SECONDARY OUTCOMES:
Visual Analogue Scale(VAS) | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  The VAS scoring system is a standardized subjective symptom assessment tool designed based on the principle of visual simulation, with a core form of a 10 cm long straight line, with a minimum score of 0 (representing no symptoms) and a maximum value of 10 (representing the most severe symptoms), with higher scores indicating more severe symptoms.
Mayo Elbow Performance Score(MEPS) | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  The Mayo Elbow Performance Score (MEPS) is a standardized tool for quantitatively assessing elbow function, with a score ranging from 0-100 , with higher scores indicating better elbow joint function (e.g.≥, 90 points are "excellent", 75-89 points are "good", and 60-74 points are "acceptable", <60 points are "poor"). The scoring system is evaluated comprehensively through four core dimensions: 1. Pain (0-45 points): graded according to pain frequency and severity, no pain is a full score, and loss of mobility is 0 points; 2. Motor function (0-20 points): based on flexion and extension mobility (20 points are scored for 100° of motion arc≥ only 5 points are scored for 50° of <); 3. Stability (0-10 points): evaluate the degree of varus laxity (no full score for relaxation, 0 points for obvious instability); 4. Daily living ability (0-25 points): Test five actions (combing hair, eating, personal hygiene, wearing shirts, shoes), 5 points for each item.
Oxford Elbow Score(OES) | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  The Oxford Elbow Score (OES) is a self-rated standardized instrument for assessing elbow disease or postoperative functional recovery on a scale of 0-100, with higher scores indicating better elbow function (e.g., better pain control, mobility, and quality of life). The scoring system consists of three aspects: 1. Elbow pain (4 questions, assessing pain frequency, intensity and impact on life); 2. Elbow function (4 questions, test mobility, grasp and daily activities); 3. Psychosocial impact (4 questions, focusing on social, emotional and appearance satisfaction).
Disabilities of the Arm, Shoulder and Hand(DASH) | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  The DASH scoring system is a standardized self-assessment tool for quantifying the assessment of upper extremity dysfunction on a scale of 0-100, with higher scores indicating more severe upper limb dysfunction (e.g., pain, limited mobility, and more significant impact on life). The scale consists of 30 core questions covering two main areas:1. Functional disability (21 questions): Evaluate daily living ability (such as opening doors, lifting objects, writing, dressing); 2. Symptoms and social impact (9 questions): quantify pain, numbness, sleep disturbance, and social/work limitations.
Range of motion | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  Normal mobility is the basis for maintaining daily movements, and restriction or excessive can lead to functional impairment. Elbow range of motion is divided into four directions, as follows: flexion, extension, pronation, and supination
Rate of Complications | Preoperatively, 1st week, 1st month, 3rd month, and 6th month postoperatively
  Rate of postoperative complications in each group, such as infection, hematoma, severe pain, joint adhesions, nerve damage, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This study will share the medical history and physical examination, imaging data (X-ray, CT, MRI, etc.) , functional scores, laboratory test results and complications of the two groups of patients with elbow cartilage defect.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Shetty AA, Kim SJ, Bilagi P, Stelzeneder D. Autologous collagen-induced chondrogenesis: single-stage arthroscopic cartilage repair technique. Orthopedics. 2013 May;36(5):e648-52. doi: 10.3928/01477447-20130426-30. PMID 23672920
- [Background] Shetty AA, Kim SJ, Shetty V, Jang JD, Huh SW, Lee DH. Autologous collagen induced chondrogenesis (ACIC: Shetty-Kim technique) - A matrix based acellular single stage arthroscopic cartilage repair technique. J Clin Orthop Trauma. 2016 Jul-Sep;7(3):164-9. doi: 10.1016/j.jcot.2016.05.003. Epub 2016 Jun 14. PMID 27489411
- [Background] Kim SJ, Shetty AA, Kurian NM, Ahmed S, Shetty N, Stelzeneder D, Shin YW, Cho YJ, Lee SH. Articular cartilage repair using autologous collagen-induced chondrogenesis (ACIC): a pragmatic and cost-effective enhancement of a traditional technique. Knee Surg Sports Traumatol Arthrosc. 2020 Aug;28(8):2598-2603. doi: 10.1007/s00167-020-05884-y. Epub 2020 Feb 17. PMID 32064573
- [Background] Jeong IH, Shetty AA, Kim SJ, Jang JD, Kim YJ, Chung YG, Choi NY, Liu CH. Autologous collagen-induced chondrogenesis using fibrin and atelocollagen mixture. Cells Tissues Organs. 2013;198(4):278-88. doi: 10.1159/000356488. Epub 2013 Dec 20. PMID 24356241